CLINICAL TRIAL: NCT06806202
Title: Comparative Evaluation of Anesthetic Efficacy of Warm and Conventional 2% Lignocaine for the Success of Inferior Alveolar Nerve Block (IANB) in Mandibular Permanent Molars: A Randomized Controlled Clinical Trial
Brief Title: Warm Versus Conventional 2% Lignocaine for IANB Efficacy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Kanza Zafar, Dr. Kanza Zafar, Principal Investigator and Resident Operative Dentistry and Endodontics, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lignocaine Efficacy in IANB
Record Dates: First submitted 2024-12-15; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Success of Inferior Alveolar Nerve Block; Inferior Alveolar Nerve Block
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- conventional (Active Comparator): Group 1: Patients receive conventional 2% lignocaine at room temperature.
  Interventions: Drug: conventional 2% lignocaine at room temperature
- warm (42 celsius) (Active Comparator): Group 2: Patients receive pre-warmed 2% lignocaine at 42°C
  Interventions: Drug: pre-warmed 2% lignocaine at 42°C

INTERVENTIONS:
Drug: conventional 2% lignocaine at room temperature — This study aims to compare the effectiveness of warm 2% lignocaine (lidocaine) versus conventional room temperature 2% lignocaine for achieving successful inferior alveolar nerve blocks (IANB) in mandibular permanent molars
  Arms: conventional
Drug: pre-warmed 2% lignocaine at 42°C — This study aims to compare the effectiveness of warm 2% lignocaine (lidocaine) versus conventional room temperature 2% lignocaine for achieving successful inferior alveolar nerve blocks (IANB) in mandibular permanent molars
  Arms: warm (42 celsius)

SUMMARY:
The study compares the anesthetic efficacy of warm versus conventional 2% lignocaine for inferior alveolar nerve block in mandibular molars, evaluating success rates and onset time.

DETAILED DESCRIPTION:
The study will be conducted following approval from the Institutional Ethics Review Committee, AFID (ANX "A"). A total of 200 eligible patients visiting the Operative Dentistry Department at the Armed Forces Institute of Dentistry will be invited to participate. The procedure will be explained to the patients in Urdu, and written informed consent will be obtained (ANX "B").

Patients will be screened for eligibility through medical history, clinical examination, necessary tests, and peri-apical radiographs. Those meeting the inclusion criteria will be randomly assigned to one of two groups using a scientific random number table.

Group 1: Patients will receive conventional 2% lignocaine (at room temperature).

Group 2: Patients will receive pre-warmed 2% lignocaine (at 42°C). Root canal treatment will begin after the inferior alveolar nerve block (IANB) is administered. 1.8 mL of the local anesthetic will be delivered over 60 seconds using a 27-gauge needle. The first investigator will randomize participants by having them choose one of two differently colored balls to determine which anesthetic preparation (conventional or pre-warmed) they will receive. The conventional 2% lignocaine will be commercially available 2% lignocaine hydrochloride with 1:200,000 epinephrine, while the pre-warmed solution will be heated in a thermostatically controlled water bath or feeder bottle warmer (Philips AVENT) to 42°C.

The second investigator, who will be blinded to group allocation, will evaluate pain immediately after the block is administered by asking patients to rate their discomfort on a Visual Analog Scale (VAS). The onset of anesthesia will also be measured by performing gingival probing every 15 seconds. After rubber dam isolation, access cavity preparation will be performed, and pulp therapy will be initiated by the first investigator. The pulp therapy will be completed as needed, and the teeth will be restored with light-cured composite resin.

ELIGIBILITY:
Inclusion Criteria:

* Permanent teeth with acutely inflamed pulp without swelling or draining sinus.
* Patient who have carious mandibular molars.
* Patients of either gender aged between 18-50 years old.
* Systemically healthy patients.
* Patients who agree to attend for recall appointments and provide a written consent

Exclusion Criteria:

* Patients on preoperative analgesics and antibiotics.
* Teeth with calcified canals and previously treated teeth.
* Pregnant and lactating mothers.
* Patients who are immunocompromised, anxious and mentally handicapped.
* Patients who are allergic to lignocaine.
* Non-vital or necrosed teeth.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Pain during administration of injection | 60 seconds
  Pain during administration of injection with 2% conventional and warm lignocaine on visual analogue scale is assessed. Visual Analog Scale, which is a tool used to measure a patient's perception of pain. It typically consists of a line, often 10 cm long, where one end represents "no pain" and the other end represents "worst possible pain." The patient marks a point on the line that corresponds to their level of pain. The distance from the "no pain" end to the point marked by the patient is then measured, usually in centimeters or millimeters, to quantify the pain intensity. Visual Analog Scale is commonly used in clinical trials to assess pain during and after procedures, as it provides a simple and reliable method for evaluating pain intensity.
Onset of anesthesia in seconds | Every 15 seconds till patient reports no sensation after stimulus (assessed up to 15 minutes after anesthesia application)
  It will be measured by gingival probing every 15 seconds till patient reports no sensation after stimulus (assessed up to 15 minutes after anesthesia application) It will be done by using both conventional and warm 2% lignocaine.

CONTACTS AND LOCATIONS:
Overall Officials: Kanza Ali Zafar, BDS, Principal Investigator — AFID
Locations (1):
- Armed Forces Institute Of Dentistry, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No